CLINICAL TRIAL: NCT02980913
Title: Difference in the Frequency of Use of Lachrymal Substitutes in Patients With Moderate to Severe Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LT 2258-PIV-05/15
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Patients with dry eye syndrome 1 (Experimental): 20 patients with dry eye syndrome, they will receive intervention 1 for one week and then cross over to intervention 2
  Interventions: Device: Thealoz Duo eye drops and Thealoz Duo gel; Device: Thealoz Duo gel
- Experimental: Patients with dry eye syndrome 2 (Experimental): 20 patients with dry eye syndrome, they will receive intervention 2 for one week and then cross over to intervention 1
  Interventions: Device: Thealoz Duo eye drops and Thealoz Duo gel; Device: Thealoz Duo gel

INTERVENTIONS:
Device: Thealoz Duo eye drops and Thealoz Duo gel — Thealoz Duo eye drops during the day + Thealoz Duo gel at night (1 drop before going to bed) for 7 days
  Other Names: Intervention 1
Device: Thealoz Duo gel — Thealoz Duo gel during the day and at night for 7 days
  Other Names: Intervention 2

SUMMARY:
Dry eye syndrome is a highly prevalent ocular disease with an increasing incidence in the elderly population.

Topically administered lubricants are the basis for treatment of this disease. Relief of symptoms in patients with moderate to severe dry eye disease is usually reached by the use of artificial tears during the day. Nighttime relief is often achieved by substances known to be more adhesive to the ocular surface, such as gels.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged over 18 years
2. Signed and dated written informed consent.
3. History of dry eye syndrome for at least 3 months
4. Tear Break Up Time (BUT) ≤ 10 seconds or Schirmer I test ≤ 5 mm and ≥ 2mm
5. OSDI ≥ 22
6. Normal ophthalmic findings except dry eye syndrome
7. No administration of topical lubricants 24 hours before the screening examination

Exclusion Criteria:

1. Presence of an ocular pathology judged by the investigator as incompatible with the study.
2. Any other clinical relevant ocular abnormality except DES.
3. History of allergy, known hypersensitivity to one of the components: the administered medical device product, fluorescein or lissamine green
4. History of known clinically relevant allergy
5. Medical or surgical history judged by the investigator to be incompatible with the study participation (hepatic or renal insufficiency; all chronic severe organic disease: metabolic, endocrine, neoplasic, hematological disease; severe psychiatric illness, etc.).
6. History of a recent acute illness with a recovery period within the 2 weeks before the inclusion visit (Day 0).
7. Pregnancy, lactation.
8. Pre-menopausal woman who is not using a reliable birth control method (oral contraceptives or coil) or is not surgically sterilized.
9. Participation in any high-speed or water-sports during the study without ocular protection (goggles or glasses).
10. Subject unable to understand the study instructions or unlikely to comply with the study schedule and treatment.
11. Participation in another clinical study in the 4 weeks before the start of the present study or at the same time as the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-05-17 (Actual)

PRIMARY OUTCOMES:
Number of drops of Thealoz Duo® eye drops and Thealoz Duo® gel instilled during the day (patient diary) | 4 weeks
  Number of drops of Thealoz Duo® eye drops and Thealoz Duo® gel instilled during the day during the observation period of one week for each medical device (patient diary)

SECONDARY OUTCOMES:
Tear Break Up Time (BUT) | 4 weeks
Schirmer I test | 4 weeks
Conjunctival and corneal staining | 4 weeks
OSDI questionnaire | 4 weeks
Quality of life of patients (VAS) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Fondi K, Wozniak PA, Schmidl D, Bata AM, Witkowska KJ, Popa-Cherecheanu A, Schmetterer L, Garhofer G. Effect of Hyaluronic Acid/Trehalose in Two Different Formulations on Signs and Symptoms in Patients with Moderate to Severe Dry Eye Disease. J Ophthalmol. 2018 Aug 1;2018:4691417. doi: 10.1155/2018/4691417. eCollection 2018. PMID 30155282